CLINICAL TRIAL: NCT02751593
Title: Thrombocytopenia in Gestational Period
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pregnancy and thrombocytopenia
Record Dates: First submitted 2016-04-17; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Immune Thrombocytopenia; Pregnancy
Keywords: pregnancy; Immune Thrombocytopenia; dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexamethasone (Experimental): dexamethasone 40mg/d for 4 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone 40mg/d for 4 days

SUMMARY:
The project was undertaking by Peking University People's Hospital and other well-known hospitals in China. Aims at evaluating efficacy and safety of dexamethasone in management of ITP in pregnancy.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, open-labeled, pilot study of 50 ITP patients in pregnancy from Peking University People's Hospital and other well-known hospitals in China. ITP patients in pregnancy who failed to respond to prednisone, IVIG and developed refractoriness to platelet transfusion will be given dexamethasone intravenously at a dose of 40mg every day for four days. Platelet count, bleeding and other symptoms will be evaluated before and after treatment. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 20-50 years old.
* After 12 weeks gestation.
* Diagnosed with ITP meeting the diagnostic criteria for immune thrombocytopenia.
* Patients who have no response or relapsed after Corticosteroid or IVIG.
* Patients developed refractoriness to platelet transfusion.
* To show a platelet count < 30×10^9/L, and with bleeding manifestations.
* Willing and able to sign written informed consent.

Exclusion Criteria:

* Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
* Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit.
* Current HIV infection or hepatitis B virus or hepatitis C virus infections.
* Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP.
* Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia).
* Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
* Patients who are deemed unsuitable for the study by the investigator.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Response rate (CR+R) | 3 months

SECONDARY OUTCOMES:
Platelet count | 2 years
Adverse events | 2 years
live birth rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-hui Zhang, Dr, Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided